CLINICAL TRIAL: NCT00065026
Title: Environmental Approaches to Reducing Obesity: Increasing Physical Activity Levels in Low-Income Women
Brief Title: Increasing Physical Activity Levels in Low-Income Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Allocation: Non-Randomized | Masking: None | Purpose: Prevention
Other Study IDs: IPALLW (completed)
Record Dates: First submitted 2003-07-16; First posted 2003-07-18 (Estimated); Last update posted 2010-01-13 (Estimated); Status verified 2010-01

CONDITIONS: Healthy

INTERVENTIONS:
Behavioral: Physical activity opportunities for low-income women

SUMMARY:
Regular physical activity is important for good health. Women, particularly women with low incomes, have many personal barriers to regular physical activity. The purpose of this study is to reduce environmental barriers to physical activity for women in two specific low-income neighborhoods (in Louisville, KY) by providing opportunities for safe physical activity and addressing barriers such as lack of child care. Two groups of women will have pretest information (cholesterol, blood sugar, blood pressure, percent body fat, height, weight, waist and hip measurements) collected and the same information 6 months later at post-test. One group will have access to multiple physical activity opportunities in their neighborhood and at the neighborhood community center. An advanced registered nurse practitioner will facilitate the activity opportunities. The groups will be compared on their pretest and post-test information to see if the group with the physical activity opportunities has increased physical activity as measured by pedometer and self-report questionnaire, and to see if there are changes in the measures tested at pre and post (measures that may be improved by regular physical activity).

ELIGIBILITY:
live in one of two specific low-income neighborhoods in Louisville, KY

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2003-04

CONTACTS AND LOCATIONS:
Locations (1):
- University of Louisville, Louisville, Kentucky, United States